CLINICAL TRIAL: NCT06883474
Title: Osteosclerotic Changes on Computed Tomography Predict Disease Progression and Poor Survival in Prostate Cancer
Brief Title: Osteosclerotic Changes on CT Predict Survival in Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Meiting Chen, Doctor, Sun Yat-sen University
Other Study IDs: SYSUCC-BONE
Record Dates: First submitted 2025-03-13; First posted 2025-03-19 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2024-10

CONDITIONS: Prostate Cancer (Adenocarcinoma); Prostate Cancer Metastatic Disease
Keywords: Bone metastasis; computed tomography; osteosclerotic change; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Osteosclerotic Changes on Computed Tomography — Osteosclerotic Changes on Computed Tomography

SUMMARY:
The study specifically investigated PC patients with bone metastasis and conducted a comprehensive analysis of the correlation between OCs and patient survival outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 1）Histopathological confirmation of prostate adenocarcinoma
* 2）Radiologically verified bone metastasis, assessed through bone scintigraphy and CT imaging from the initiation of systemic therapy until disease progression.

Exclusion Criteria:

* 1）Lacking of complete clinical profiles.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Prostate cancer patients with bone metastasis
Sampling Method: Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2010-07-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Radiographic progression-free survival | From enrollment to the end of treatment at 5 years

SECONDARY OUTCOMES:
overall survival | From enrollment to the end of treatment at 5 years

IPD SHARING:
Plan to Share IPD: No